CLINICAL TRIAL: NCT02772965
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Pragmatic Clinical Trial To Evaluate The Effectiveness Of Low Dose Oral Methotrexate In Patients With Pediatric Crohn's Disease Initiating Anti-TNF Therapy
Brief Title: Low Dose Oral Methotrexate in Pediatric Crohn's Disease Patients Initiating Anti-Tumor Necrosis Factor (Anti-TNF) Therapy
Acronym: COMBINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); ImproveCareNow (ICN) (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); Children's Hospital Medical Center, Cincinnati (Other); Grifols Diagnostics Solutions, Inc (Unknown); National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-0476; PCS-1406-18643 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI)); 1U19AR069525-01 (NIH); PCD-MTX-001 (Other: UNC)
Record Dates: First submitted 2016-04-27; First posted 2016-05-16 (Estimated); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-06

CONDITIONS: Pediatric Crohn's Disease
MeSH Terms: conditions — Pediatric Crohn's disease | interventions — Methotrexate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Experimental): Methotrexate (10, 12.5, or 15 mg), once weekly. Weight-based dosing. Ondansetron (4 mg), twice weekly, 1 hour prior to methotrexate dose and the morning after methotrexate dose.
  Folic Acid (1 mg) daily
  Interventions: Drug: Methotrexate
- Sugar pill (placebo) (Placebo Comparator): Placebo for methotrexate, once weekly. Placebo for ondansetron, twice weekly, 1 hour prior to methotrexate placebo dose and the morning after methotrexate placebo dose.
  Folic Acid (1 mg) daily
  Interventions: Other: Sugar pill (placebo)

INTERVENTIONS:
Drug: Methotrexate — 1. Oral methotrexate (MTX): The weekly dose will be 15 mg for children ≥ 40kg, 12.5 mg for children 30 to <40 kg, and 10 mg for children 20 to <30 kg.
  2. A twice per week, 4mg dose of ondansetron will be provided as pre-treatment to prevent nausea (study provider may opt-out of this component based on clinical judgement).
  3. A 1 mg dose of folic acid per day will be provided. This will help to reduce the risk of side effects in the MTX group.
  Drug kits will contain a 3 month supply of each medication. Refills will be provided every 3 months until week 156 unless there is a failure to induce and maintain remission, development of unacceptable toxicity, pregnancy in a female participant, or failure of the participant to attend scheduled study visits.
  Other Names: Methotrexate Sodium
  Arms: Methotrexate
Other: Sugar pill (placebo) — 1. Placebo for methotrexate: The weekly dose will mimic that of methotrexate.
  2. Placebo for ondansetron: The weekly dose will mimic that of ondansetron (study provider may opt-out of this component based on clinical judgement).
  3. A 1 mg dose of folic acid per day will be provided to maintain blinding.
  Drug kits will contain a 3 month supply of each medication. Refills will be provided every 3 months until week 156 unless there is a failure to induce and maintain remission, development of unacceptable toxicity, pregnancy in a female participant, or failure of the participant to attend scheduled study visits.
  Arms: Sugar pill (placebo)

SUMMARY:
The purpose of this study is to determine whether adding low dose methotrexate to anti -TNF therapy is more effective than treatment with anti-TNF therapy alone in inducing and maintaining steroid-free remission for children with Crohn's Disease.

DETAILED DESCRIPTION:
Overall study duration: 6 years Multi-center study: up to 42 centers

Number of subjects: 425 Duration of treatment for each subject: up to 156 weeks (3 years)

The primary endpoint is percent of patients who experienced treatment failure over time.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Crohn's Disease (PCD) patients, < 21 years of age, ≥20 kg, initiating anti-TNF therapy with infliximab or adalimumab (including biosimilars).
* Diagnosis of Crohn's Disease (CD) established confirmed by the treating clinician, and established by standard clinical criteria (radiography, endoscopy, histology).
* Ability to provide parental permission and child assent (where applicable), or adult consent for patients ages 18-20.

Exclusion Criteria:

* Prior use of anti-TNF or other biological therapy for CD
* Lack of stable home address that study medications can be mailed to
* Anticipated short length of follow up at study center (plans for family to move, transition to adult GI (gastrointestinal) provider, etc.). Patients expected to leave practice < 12 months from enrollment should not be enrolled.
* Concurrent pelvic or abdominal abscess. A recent history of abdominal or pelvic abscess, which is controlled, does not exclude the subject.
* Prior intra-abdominal surgery without a clinically significant relapse (i.e. patients starting on anti-TNF for post-op prophylaxis or for endoscopic recurrence only should not be included)
* Receipt of a live virus vaccine within the last 30 days
* Pregnancy, planning to become pregnant, or high risk of pregnancy as determined by the local investigator
* Breastfeeding
* Refusal to stay abstinent or utilize 2 forms of birth control while on study medication (for female patients)
* BMI > 98% for gender and age
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years). A recent history of basal cell or squamous cell carcinoma, which is considered surgically cured, does not exclude the subject.Those with a recent history of colonic adenoma or dysplastic lesions should be excluded.
* Known high alcohol consumption (more than seven drinks per week)
* Patients with serum albumin < 2.5 g/dl
* Patients with white blood cell count (WBC) < 3.0 x109th/L
* Patients with platelet count < 100 x109th/L
* Patients with initial elevation of liver enzymes (AST or ALT) > 1.5 times above normal limit
* Patients with known active infection with Clostridium difficile (C. difficile) (untreated infection based on clinician assessment does not apply to colonization or infection controlled with current or prior treatment.)
* Patients with pre-existing hepatic disease
* Patients with pre-existing renal dysfunction (creatinine > 0.8 for children age<10, creatinine > 1.2 mg/dl for children age 10-18, and creatinine > 1.5 mg/dl for adults age 18 years and older).
* Patients with a pre-existing chronic lung disease other than well controlled asthma
* Current treatment with one of the following drugs: Probenecid (Probalan), Acitretin (Soriatane), Streptozocin (Zanosar), Azathioprine (Imuran, Azasan), 6-mercaptopurine (Purinethol, Purixan)
* Other concerns about the patient/family's ability to participate in the study

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 306 (Actual)
Dates: Start 2016-10; Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Kappelman, MD, Study Director — University of North Carolina, Chapel Hill
Locations (32):
- United States (32):
  - Children's of Alabama, Birmingham, Alabama
  - Stanford Children's Health, Alto, California
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Nemours Children's Health System - Wilmington, Wilmington, Delaware
  - Nemours Children's Health System - Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Health System - Orlando, Orlando, Florida
  - Children's Healthcare of Atlanta at Egleston/Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - MassGeneral Hospital for Children, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan | CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - St. Louis Children's Hospital | Washington University, St Louis, Missouri
  - Children's Hospital and Medical Center Omaha, Omaha, Nebraska
  - Mount Sinai Kravis Children's Hospital, New York, New York
  - Upstate Golisano Children's Hospital, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - The University of Vermont Children's Hospital, Burlington, Vermont
  - Pediatric Specialists of Virginia, Fairfax, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kappelman MD, Wohl DA, Herfarth HH, Firestine AM, Adler J, Ammoury RF, Aronow JE, Bass DM, Bass JA, Benkov K, Tobi CB, Boccieri ME, Boyle BM, Brinkman WB, Cabera JM, Chun K, Colletti RB, Dodds CM, Dorsey JM, Ebach DR, Entrena E, Forrest CB, Galanko JA, Grunow JE, Gulati AS, Ivanova A, Jester TW, Kaplan JL, Kugathasan S, Kusek ME, Leibowitz IH, Linville TM, Lipstein EA, Margolis PA, Minar P, Molle-Rios Z, Moses J, Olano KK, Osaba L, Palomo PJ, Pappa H, Park KT, Pashankar DS, Pitch L, Robinson M, Samson CM, Sandberg KC, Schuchard JR, Seid M, Shelly KA, Steiner SJ, Strople JA, Sullivan JS, Tung J, Wali P, Zikry M, Weinberger M, Saeed SA, Bousvaros A. Comparative Effectiveness of Anti-TNF in Combination With Low-Dose Methotrexate vs Anti-TNF Monotherapy in Pediatric Crohn's Disease: A Pragmatic Randomized Trial. Gastroenterology. 2023 Jul;165(1):149-161.e7. doi: 10.1053/j.gastro.2023.03.224. Epub 2023 Mar 31. PMID 37004887

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate: Methotrexate (10, 12.5, or 15 mg), once weekly. Weight-based dosing. Ondansetron (4 mg), twice weekly, 1 hour prior to methotrexate dose and the morning after methotrexate dose.
  Folic Acid (1 mg) daily
  Methotrexate: 1) Oral methotrexate (MTX): The weekly dose will be 15 mg for children ≥ 40kg, 12.5 mg for children 30 to <40 kg, and 10 mg for children 20 to <30 kg. 2) A twice per week, 4mg dose of ondansetron will be provided as pre-treatment to prevent nausea (study provider may opt-out of this component based on clinical judgement). 3) A 1 mg dose of folic acid per day will be provided. This will help to reduce the risk of side effects in the MTX group.
  Drug kits will contain a 3 month supply of each medication. Refills will be provided every 3 months until week 156 unless there is a failure to induce and maintain remission, development of unacceptable toxicity, pregnancy in a female participant, or failure of the participant to attend scheduled study visits.
- Sugar Pill (Placebo): Placebo for methotrexate, once weekly. Placebo for ondansetron, twice weekly, 1 hour prior to methotrexate placebo dose and the morning after methotrexate placebo dose.
  Folic Acid (1 mg) daily
  Sugar pill (placebo): 1) Placebo for methotrexate: The weekly dose will mimic that of methotrexate. 2) Placebo for ondansetron: The weekly dose will mimic that of ondansetron (study provider may opt-out of this component based on clinical judgement). 3) A 1 mg dose of folic acid per day will be provided to maintain blinding.
  Drug kits will contain a 3 month supply of each medication. Refills will be provided every 3 months until week 156 unless there is a failure to induce and maintain remission, development of unacceptable toxicity, pregnancy in a female participant, or failure of the participant to attend scheduled study visits.
Period: Overall Study
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Started | 162 | 144
Randomized | 162 | 144
Withdrew Before Receiving Drug | 6 | 3
Modified Intent to Treat | 156 | 141
Completed | 140 | 126
Not Completed | 22 | 18

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat population presented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Sugar Pill (Placebo) | Total
Number analyzed (Participants) | 156 | 141 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (2.5) | 14.0 (2.8) | 13.9 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 104
  Male | 103 | 90 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 150 | 138 | 288
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 19 | 32
  White | 131 | 113 | 244
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 156 | 141 | 297
Tumor Necrosis Factor (TNF) Inhibitor at Baseline [Count of Participants; unit: Participants]
  Infliximab | 110 | 102 | 212
  Adalimumab | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Experiencing Treatment Failure
Description: Treatment failure is defined as follows:
  1. Failure to achieve remission (short pediatric Crohn's disease activity index [SPCDAI] < 15) by the week 26 visit;
  2. If study initiated on steroids, failure to complete steroid taper by week 16;
  3. Short pediatric Crohn's disease activity index (SPCDAI) ≥ 15 attributed to active Crohn's disease, at two or more consecutive visits beyond the week 26 visit. Elevated SPCDAI (≥ 15) due to a non-Inflammatory Bowel Disease (IBD) reason does not count toward this outcome;
  4. Hospitalization for active Inflammatory Bowel Disease or abdominal surgery after week 25;
  5. Use of oral prednisone or prednisolone, enteral release budesonide, or intravenous (IV) methylprednisolone for over 10 weeks cumulatively, beyond week 16;
  6. Discontinuation of anti-TNF agent and/or study drug for lack of effectiveness or toxicity.
Time Frame: From randomization until treatment failure, assessed up to 3 years.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Number analyzed (Participants) | 156 | 141
percentage of participants | 25.64 | 34.04
Statistical Analysis 1: Comparison: Methotrexate vs Sugar Pill (Placebo); Test type: Superiority; p = 0.08, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.45 to 1.05]

2. Secondary Outcome: Mean Patient Reported Outcome Measurement and Information System (PROMIS ) Pain Interference T-score-52 Weeks
Description: T-scores are a continuous variable. The mean in the general population is 50 (SD=10). Scores above 50 represent higher than average pain interference and scores below 50 represent lower than average pain interference. Minimal important differences (MIDs) for many PROMIS domains are in the range of 2 to 6.
  The investigators will compare the mean of PROMIS Pain Interference T-scores at week 52 between the treatment groups.
Time Frame: Weeks 52 from randomization
Population: Population includes those who completed surveys.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Number analyzed (Participants) | 119 | 107
T-score | 37.5 (12.0) | 39.5 (11.9)
Statistical Analysis 1: Comparison: Methotrexate vs Sugar Pill (Placebo); Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, Standard Error of Mean 1.4

3. Secondary Outcome: Mean Patient Reported Outcome Measurement and Information System (PROMIS ) Pain Interference T-score-week 104
Description: T-scores are a continuous variable. The mean in the general population is 50 (SD=10). Scores above 50 represent higher than average pain interference and scores below 50 represent lower than average pain interference. Minimal important differences (MIDs) for many PROMIS domains are in the range of 2 to 6.
  The investigators will compare the mean of PROMIS Pain Interference T-scores at week 104 between the treatment groups
Time Frame: 104 weeks from randomization
Population: Population includes those who completed surveys.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Number analyzed (Participants) | 91 | 77
T-score | 38.1 (12.4) | 39.9 (13.5)
Statistical Analysis 1: Comparison: Methotrexate vs Sugar Pill (Placebo); Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, Standard Error of Mean 1.8

4. Secondary Outcome: Mean PROMIS (Patient Reported Outcome Measurement and Information System) Fatigue T Score-week 52
Description: T-scores are a continuous variable. The mean in the general population is 50 (SD=10). Scores above 50 represent higher than average fatigue and scores below 50 represent lower than average fatigue. Minimal important differences (MIDs) for many PROMIS domains are in the range of 2 to 6.
  The investigators will compare the mean of PROMIS Fatigue T-scores at week 52 between the treatment groups
Time Frame: Week 52 from randomization
Population: Population includes those who completed surveys.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Number analyzed (Participants) | 119 | 107
T-score | 41.8 (14.4) | 41.8 (14.0)
Statistical Analysis 1: Comparison: Methotrexate vs Sugar Pill (Placebo); Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, Standard Error of Mean 1.6

5. Secondary Outcome: Mean PROMIS (Patient Reported Outcome Measurement and Information System) Fatigue T Score-week 104
Description: T-scores are a continuous variable. The mean in the general population is 50 (SD=10). Scores above 50 represent higher than average fatigue and scores below 50 represent lower than average fatigue. Minimal important differences (MIDs) for many PROMIS domains are in the range of 2 to 6.
  The investigators will compare the mean of PROMIS Fatigue T-scores at week 104 between the treatment groups
Time Frame: 104 weeks from randomization
Population: Population includes those who completed surveys.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Number analyzed (Participants) | 91 | 77
T-score | 41.1 (14.5) | 41.5 (14.9)
Statistical Analysis 1: Comparison: Methotrexate vs Sugar Pill (Placebo); Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Final Values) = 0.9, Standard Error of Mean 1.9

6. Secondary Outcome: Percent of Patients With Positive Anti-TNF Antibody
Description: Percent of patients with positive anti-TNF antibody will be compared between the two treatment groups using the chi-squared test.
Time Frame: Between 6 months and 2 years from randomization
Population: Analysis includes participants who provided a blood sample.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Sugar Pill (Placebo)
Number analyzed (Participants) | 112 | 100
percentage of participants | 28.5 | 40
Statistical Analysis 1: Comparison: Methotrexate vs Sugar Pill (Placebo); Test type: Superiority; p = 0.08, Chi-squared; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.49 to 1.04]

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent until study completion, up to 3 years.
Arm/Group | Methotrexate | Sugar Pill (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/141
Serious Adverse Events (participants affected / at risk) | 23/156 | 28/141
Other Adverse Events (participants affected / at risk) | 156/156 | 129/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Methotrexate (N=156) | Sugar Pill (Placebo) (N=141)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 7 (8)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease exacerbation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
G-Tube placement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileocecectomy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3/3 (3) | 2 (2)
Perirectal abscess (Gastrointestinal disorders) | 1 (1) | 1 (1)
post-operative infection from ileocecectomy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis - right ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Nervous system disorders) | 1 (1) | 0 (0)
Other Paranoia and mental status change (Psychiatric disorders) | 0 (0) | 1 (1)
Severe major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 3 (3) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 2 (2)
cervical lymphodenitis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute cellutis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anti-TNF Infusion related reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Facial abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Facial flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tonsillectomy and adenoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=156) | Sugar Pill (Placebo) (N=141)
Nausea (Gastrointestinal disorders) | 32 (38) | 19 (30)
Abdominal Discomfort (Gastrointestinal disorders) | 23 (35) | 17 (23)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 12 (15)
Elevation of Liver Enzymes (AST, ALT) (Hepatobiliary disorders) | 20 (22) | 8 (9)
Fever (General disorders) | 11 (12) | 8 (9)
Fatigue (General disorders) | 8 (11) | 9 (12)
Headache (Nervous system disorders) | 12 (13) | 18 (20)
Rash (Skin and subcutaneous tissue disorders) | 17 (22) | 17 (20)
C. Difficile (Infections and infestations) | 8 (10) | 7 (10)
Strep pharyngitis (Infections and infestations) | 10 (13) | 6 (7)
Upper Respiratory Infection (Infections and infestations) | 8 (9) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02772965/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT02772965/SAP_001.pdf